CLINICAL TRIAL: NCT04987528
Title: Incidence, Risk Factors and Prognosis of Pulmonary Fibrosis During Severe COVID-19 Pneumonia
Brief Title: Pulmonary Fibrosis During Severe COVID-19 Pneumonia
Acronym: FIBRO-COVID
Status: Active, not recruiting | Type: Observational
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021_06_02_JAS
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2; Acute Respiratory Distress Syndrome; Pulmonary Fibrosis
Keywords: Mechanical Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pulmonary fibrosis: All ICU patients for which one of the non-invasive criteria of pulmonary fibrosis is reached :
  * Typical CT scan patterns (reticulation and/or bronchiectasia)
  * Serum PIIINP above 16 µg/L
  * BAL PIIINP above 9 µg/L
  Interventions: Diagnostic Test: Aminoterminal type III peptide of procollagen; Diagnostic Test: Lung computed tomography
- Patients without pulmonary fibrosis: All ICU patients for which none of the non-invasive criteria of pulmonary fibrosis are reached.
  Interventions: Diagnostic Test: Aminoterminal type III peptide of procollagen; Diagnostic Test: Lung computed tomography

INTERVENTIONS:
Diagnostic Test: Aminoterminal type III peptide of procollagen — Serial Measurement of PIIINP in serum and/or BAL
  Other Names: PIIINP
Diagnostic Test: Lung computed tomography — Screening for the presence of reticulation or bronchiectasia within lung parenchyma
  Other Names: Chest CT scan

SUMMARY:
The COVID-19 pandemic is caused by the severe acute respiratory syndrome coronavirus 2 (SARS CoV-2), an emerging coronavirus, which has already infected 192 million people with a case fatality rate close to 2%. About 5% of patients infected with SARS CoV-2 have a critical form with organ failure. Among critical patients admitted to intensive care, about 70% of them will require ventilatory assistance by invasive mechanical ventilation (MV) with a mortality rate of 35% and a median MV duration of 12 days. The most severe lung damage resulting from SARS CoV-2 infection is the acute respiratory distress syndrome (ARDS). The virus infects alveolar epithelial cells and capillary endothelial cells leading to an activation of endothelium, hypercoagulability and thrombosis of pulmonary capillaries. This results in abnormal ventilation / perfusion ratios and profound hypoxemia. To date, the therapeutic management of severe SARS CoV-2 pneumonia lay on the early use of corticosteroids and Interleukin-6 (IL-6) receptor antagonist, which both reduce the need of MV and mortality. The risk factors of death in Intensive Care Unit (ICU) are: advanced age, severe obesity, coronary heart disease, active cancer, severe hypoxemia, and hepatic and renal failure on admission. Among MV patients, the death rate is doubled in those with both reduced thoracopulmonary compliance and elevated D-dimer levels. Patients with severe alveolar damage are at risk of progressing towards irreversible pulmonary fibrosis, the incidence of which still remain unknown. The diagnosis of pulmonary fibrosis is based on histology but there are some non-invasive alternative methods (serum or bronchoalveolar biomarkers, chest CT scan). We aim to assess the incidence of pulmonary fibrosis in patients with severe SARS CoV-2 related pneumonia. We will investigate the prognostic impact of fibrosis on mortality and the number of days alive free from MV at Day 90. Finally, we aim to identify risk factors of fibrosis.

DETAILED DESCRIPTION:
Medical charts of patients admitted at the Intensive Care Unit (ICU) of the European Hospital of Marseille between March 2020 and June 2021 will be collected retrospectively using electronic database. Data collected will focus on demography, clinical variables, biological analyses, lung biopsies, and chest CT scans performed during the hospital stay.

Our routine protocol for COVID-19 management follows the "Coronavirus Disease 2019 (COVID-19) Treatment Guidelines" including the early use of corticosteroids (Dexamethasone) and IL-6 receptor antagonist (Tocilizumab). Additionally, we routinely perform, on a weekly basis, measurements of SARS CoV-2 viral load by PCR, SARS CoV-2 antibodies production, and biomarkers of fibrosis including hyaluronic acid (HA) and amino-terminal type I (PINP) and type III (PIIINP) peptides of procollagen.

The present study aim to determine the proportion of patients encountering non-invasive criteria of pulmonary fibrosis as defined by either typical CT scan patterns (reticulation and/or bronchiectasia), or increased serum concentration of PIIINP above 16 µg/L, or increased bronchoalveolar lavage (BAL) concentration of PIIINP above 9 µg/L.

A definitive diagnosis of lung fibrosis will be established according to lung pathology findings in patients for whom a lung biopsy have been performed during the hospital stay.

Patients with a diagnosis of pulmonary fibrosis will be compared with those without fibrosis, both in the population of mechanically ventilated patients and in those remained spontaneously breathing.

The primary end-point will be the number of days alive and free from the ventilator (ventilator-free days) at Day 90. The others outcomes of interest will be the duration of mechanical ventilation, the duration of ICU stay, the ICU mortality, the in-hospital mortality, the Day 28 mortality, and the Day 90 mortality.

The present study also aims to determine the risk factors of pulmonary fibrosis occurence, focusing on mechanical ventilatory settings, daily dose of corticosteroids, and the occurence of nosocomial pneumonia with special attention to lung reactivation of herpesviridae.

Finally, the relation between antibodies production and viral clearance (defined as the time to the first negative SARS CoV-2 PCR) or ICU survival will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Acute hypoxemic respiratory failure
* Positive SARS CoV-2 PCR on nasopharyngeal swab or distal airway sampling
* ICU admission during the hospital stay

Exclusion Criteria:

* Chronic respiratory failure (Oxygen or NIPPV at home)
* Patients with "Do Not Resuscitate" order at ICU admission
* Admission from an other ICU with a stay > 2 days
* Transfer to an another ICU during the ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will focused on patients with severe SARS Cov-2 pneumonia requiring ICU admission.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free days | Day 90
  Number of days alive and free from mechanical ventilation

SECONDARY OUTCOMES:
Day 90 mortality | Day 90
  Mortality at Day 90
Day 28 mortality | Day 28
  Mortality at Day 28
ICU Mortality | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Death from any cause during the ICU stay
In-hospital Mortality | From date of hospital admission until the date of hospital liberation, assessed up to 12 months
  Death from any cause during the Hospital stay
Length of MV | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Duration of mechanical ventilation during the ICU stay
Length of ICU stay | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Duration of ICU stay
Length of hospital stay | From date of hospital admission until the date of hospital liberation, assessed up to 12 months
  Duration of hospital stay
Time to viral clearance | From date of first symptom until the date of ICU liberation, assessed up to 6 months
  Time from first symptom to the first negative SARS CoV-2 PCR
Corticosteroid dose | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Daily corticosteroid dose (methylprednisolone equivalent)
Lung herpesviridae reactivation | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Presence on BAL of at least one Herpesviridae (Cytomegalovirus, Epstein-Barr Virus, Herpes simplex virus, Human herpes virus-6)
Blood herpesviridae reactivation | From date of ICU admission until the date of ICU liberation, assessed up to 6 months
  Presence on serum of at least one Herpesviridae (Cytomegalovirus, Epstein-Barr Virus, Herpes simplex virus, Human herpes virus-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Europeen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] COVID-ICU Group on behalf of the REVA Network and the COVID-ICU Investigators. Clinical characteristics and day-90 outcomes of 4244 critically ill adults with COVID-19: a prospective cohort study. Intensive Care Med. 2021 Jan;47(1):60-73. doi: 10.1007/s00134-020-06294-x. Epub 2020 Oct 29. PMID 33211135
- [Background] Grasselli G, Tonetti T, Protti A, Langer T, Girardis M, Bellani G, Laffey J, Carrafiello G, Carsana L, Rizzuto C, Zanella A, Scaravilli V, Pizzilli G, Grieco DL, Di Meglio L, de Pascale G, Lanza E, Monteduro F, Zompatori M, Filippini C, Locatelli F, Cecconi M, Fumagalli R, Nava S, Vincent JL, Antonelli M, Slutsky AS, Pesenti A, Ranieri VM; collaborators. Pathophysiology of COVID-19-associated acute respiratory distress syndrome: a multicentre prospective observational study. Lancet Respir Med. 2020 Dec;8(12):1201-1208. doi: 10.1016/S2213-2600(20)30370-2. Epub 2020 Aug 27. PMID 32861276
- [Background] Forel JM, Guervilly C, Hraiech S, Voillet F, Thomas G, Somma C, Secq V, Farnarier C, Payan MJ, Donati SY, Perrin G, Trousse D, Dizier S, Chiche L, Baumstarck K, Roch A, Papazian L. Type III procollagen is a reliable marker of ARDS-associated lung fibroproliferation. Intensive Care Med. 2015 Jan;41(1):1-11. doi: 10.1007/s00134-014-3524-0. Epub 2014 Oct 30. PMID 25354475
- [Background] Burnham EL, Hyzy RC, Paine R 3rd, Kelly AM, Quint LE, Lynch D, Curran-Everett D, Moss M, Standiford TJ. Detection of fibroproliferation by chest high-resolution CT scan in resolving ARDS. Chest. 2014 Nov;146(5):1196-1204. doi: 10.1378/chest.13-2708. PMID 24722949
- See also: World Health Organization Coronavirus (COVID-19) Dashboard — https://covid19.who.int/